CLINICAL TRIAL: NCT00727116
Title: Pennsylvania Abusive Head Trauma Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Pennsylvania Department of Health (Other Government); American Academy of Pediatrics (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U49CE001274 (NIH)
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Injury; Traumatic Brain Injury; Child Abuse
MeSH Terms: conditions — Wounds and Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- State-wide (Experimental): All parents of newborns in Pennsylvania hospitals will receive the parent education materials
  Interventions: Behavioral: PA Abusive Head Trauma Prevention Program: State-wide
- Central PA (Experimental): All of Central PA new parents will receive the state-wide hospital-based intervention. In half of the 31 central PA counties, all primary care providers having offices in those counties provide an office-based booster intervention to new parents. The other half of central PA counties will receive the state-wide, hospital-based intervention, but not the office-based booster intervention.
  Interventions: Behavioral: PA Abusive Head Trauma Prevention Program: State-wide; Behavioral: PA Abusive Head Trauma Prevention Program Booster: Central PA

INTERVENTIONS:
Behavioral: PA Abusive Head Trauma Prevention Program: State-wide — Upon the birth of the child in a Pennsylvania hospital, all parents (mothers, and whenever possible, fathers or father figures) will be asked to read written materials and view an 8-minute video on the dangers of violent infant shaking. Parent education materials contain four key messages: crying is a normal infant behavior, how to keep calm when an infant is crying, how to help calm a crying infant, how to select other caregivers for your infant. Parents will be asked to voluntarily sign a commitment statement affirming their receipt and understanding of the materials.
Behavioral: PA Abusive Head Trauma Prevention Program Booster: Central PA — All primary care providers serving families of newborns in half of the counties in Central PA will be asked to provide all parents of newborns at the 2-, 4-, and 6-month immunization visits another set of written materials about violent infant shaking and voluntarily sign a response form that they read and understood the materials.
  Arms: Central PA

SUMMARY:
This project is designed to evaluate a statewide, hospital-based parent education program to prevent abusive head trauma (AHT) in Pennsylvania, and investigate the additional effectiveness and cost-effectiveness of "booster" sessions of parent education delivered to parents at primary care provider offices in central Pennsylvania.

Specific Aims:

1. Assess the effectiveness of an established statewide program of hospital-based postnatal parent education about violent infant shaking, provided at a single consistent point in time between the infant's birth and hospital discharge, in reducing the incidence of AHT.
2. Identify which component(s) are the most important mediators of the intervention's effectiveness; determine whether the intervention effect is more directly related to changes in perpetrator or caregiver behavior; and determine the effectiveness of the intervention among various socioeconomic groups.
3. Determine the cost effectiveness of the hospital-based program.
4. Establish the feasibility, additional costs, and effectiveness of a combined program of repeated exposure delivered both post-natally in the hospital and during follow up 2-, 4- and 6-month outpatient health maintenance visits with the pediatric care provider.

DETAILED DESCRIPTION:
Upon the birth of the child, all parents (mothers, and whenever possible, fathers or father figures) will be asked to read written materials and view an 8-minute video on the dangers of violent infant shaking. Parents will be asked to voluntarily sign a commitment statement affirming their receipt and understanding of the materials; these commitment statements will be sent to the Principal Investigator. A random subset of parent participants will be asked to voluntarily answer a short questionnaire about their impressions of the materials. In addition, 31 counties in central Pennsylvania will be randomly divided into two groups. In 15 counties, the hospital-based intervention will remain as described above. In the other 16 counties, all primary care providers having offices in those counties will be asked to provide all parents of newborns at the 2-, 4-, and 6-month immunization visits another set of written materials about violent infant shaking and voluntarily sign a response form that they read and understood the materials. Participating parents in this group will also be asked if they would be willing to complete a short telephone survey when the infant is 7 months old (and if so, asked to provide a telephone number). The telephone survey asks questions about the intervention materials and parents' perception of the information, and seeks to determine the mediators of a program effect. An invitation letter will be sent to a control group of parents who do not receive the office-based intervention to ask if they would be willing to complete the short telephone survey when their infant is 7 months old.

ELIGIBILITY:
Inclusion Criteria:

* Parents giving birth in a PA hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 949609 (Actual)
Dates: Start 2008-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Incidence of abusive head trauma in infants | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dias, MD, FAAP, Principal Investigator — Penn State University Hershey Medical Center

REFERENCES:
- [Background] Dias MS, Smith K, DeGuehery K, Mazur P, Li V, Shaffer ML. Preventing abusive head trauma among infants and young children: a hospital-based, parent education program. Pediatrics. 2005 Apr;115(4):e470-7. doi: 10.1542/peds.2004-1896. PMID 15805350